CLINICAL TRIAL: NCT03803735
Title: French African Pediatric Oncology Registry
Brief Title: Hospital Based Registry of Childhood Cancer in Pediatric Oncology Units in French Speaking Africa
Acronym: RFAOP
Status: Recruiting | Type: Observational
Sponsor: French Africa Pediatric Oncology Group (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: GFAOP
Record Dates: First submitted 2018-11-08; First posted 2019-01-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The ultimate aim of this registry is to collect precise information concerning the children coming to oncology units working with the French African Oncology Group. This data will help to plan and provide correct pediatric oncology treatment and care for this population.

Collecting the data will give much needed information on numbers, stage, treatment and outcome. The register will give data for local and national health authorities in planning pediatric cancer programs.

DETAILED DESCRIPTION:
This register is a registration of all children entering hospital based pediatric oncology units, working in selected hospitals in French speaking Africa. The data collected includes: demographic and socioeconomic status as well as clinical status and outcome.

The register also collects information on vital status, treatment abandonment and loss to follow-up.

Data, collected locally is entered on line using the Research Electronic Data Capture (REDCap) program. Data are stored under the responsibility of the IT department at Gustave ROUSSY in Paris- Villejuif.

ELIGIBILITY:
Inclusion Criteria:

1. Any child presenting at any one of the participating units for treatment
2. Any child with any type of cancer
3. Any child or adolescent less than 18 years of age.

Exclusion Criteria:

1. No cancer found
2. Age greater than 18 years -

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All childre with any pediatric cancer types, coming into any one of the participating units in a 12 month period.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of children with a suspicion of any type of cancer in a given unit | in any 12 month period
  Number of children with details of :
  1. the type of cancer
  2. the stage of the identified cancer coming into a given unit
VITAL STATUS: | in any 12 month period
  Dead or alive
  1. The number of children living
  2. the number of children dead
Illness status | in any 12 month period
  1. The number of children relapsed,
  2. The number of children whos illness has progressed.
Treatment Status | in any 12 month period
  1. The number of children who had treatment administered,
  2. The number of children who abandoned treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Mallon, MSc, Study Director — French Africa Pediatric Oncology Group
Locations (14):
- Burkina Faso (2):
  - Hopital Yalgado Ouedraogo, Ouagadougou
  - Centre Hospitalier Universitaire Pédiatrique Charles De Gaulle, Ouagadougou
- Centre Mère et Enfant CME-FCB (Fondation Chantal Biya), Yaoundé, Cameroon
- CHU de Treichville à ABIDJAN, Abidjan, Abidjan Autonomous District, Côte d’Ivoire
- Democratic Republic of the Congo (2):
  - Cliniques Universitaires de Kinshasa, Kinshasa, Kinshasa City
  - Cliniques Universitaires de Lubumbashi (CUL), Lubumbashi
- GFAOP, Villejuif, PARIS, France
- l'Institut de Cancérologie de Libreville, Libreville, Gabon
- HJRA, Hôpital universitaire Joseph Ravoahangy Andrianavalona, Antananarivo, Ampefiloha, Madagascar
- CHU Gabriel Touré (HGT), Bamako, Mali
- Centre National d'Oncologie (CNO), Nouakchott, Mauritania
- CNLC, Centre National de Lutte contre le Cancer, Niamey, Niger
- Hôpital Aristide Le Dantec, Avenue Pasteur, BP 3001, Dakar, Dakar, Senegal
- CHU Sylvanus Olympio, Lomé, Togo

IPD SHARING:
Plan to Share IPD: Undecided
Units have acess to their own data and can use it for reporting.